CLINICAL TRIAL: NCT01064362
Title: Risk of Hemorrhage in Patients Prescribed Arixtra Compared to LMWH
Brief Title: Hemorrhage Risk Prescribed Arixtra
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113962; EPI40612 (Other: GSK); WEUSRTP4388 (Other: GSK)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2011-06

CONDITIONS: Thrombosis, Venous
Keywords: Haemorrhage; Thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis; Hemorrhage | interventions — Fondaparinux; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prophylaxis following major orthopedic surgery: Patients age 18 years and older in the PHARMO RLS database treated with either fondaparinux sodium or LMWH for thromboprophylaxis following hip fracture and/or hip/knee replacement surgery.
  Interventions: Drug: Fondaparinux sodium; Drug: Low molecular weight heparin (LMWH)

INTERVENTIONS:
Drug: Fondaparinux sodium — Fondaparinux sodium for thromboprophylaxis (ATC: B01AX05)
Drug: Low molecular weight heparin (LMWH) — LMWH including: dalteparin, nadroparin, enoxaparin or tinzaparin (ATC:B01AB (excluding B01AB01))

SUMMARY:
Arixtra (fondaparinux sodium) was the first selective Factor Xa inhibitor to be marketed. As with all anticoagulants, an important adverse event associated with Arixtra use is haemorrhage. Previous studies using clinical trial and observational data show no difference in the risk of haemorrhage in patients treated with Arixtra compared to (low molecular weight heparins) LMWHs. This study will assess the risk of haemorrhage in major orthopaedic surgery patients (hip fracture surgery and/or hip/knee replacement surgery) treated with either Arixtra or LMWH for thromboprophylaxis and will provide additional observational data from a European country to strengthen the comprehensive review of haemorrhage and the post-marketing safety of Arixtra. All patients age 18 years and older with a primary discharge diagnosis for hip fracture surgery and/or a hospitalization for hip and/or knee replacement surgery from the PHARMO RLS database in the Netherlands are eligible for participation. For study inclusion patients must receive either Arixtra or LMWH as initial in-hospital thromboprophylactic agent and have at least three months in the PHARMO RLS database before cohort entry date. Patients with a history of hospitalization for haemorrhage, renal failure or liver failure in the past 3 months will be excluded. Descriptive statistics, including gender, age, length of treatment, co-morbidities, concomitant medications, and other covariates will be calculated.

Data for this study were obtained from different registers in the PHARMO medical record linkage system (PHARMO RLS) in the Netherlands. The PHARMO medical record linkage system is a population-based patient-centric data tracking system that includes high quality and complete information of patient demographics, drug dispensing, and hospital morbidity records of approximately 2.3 million community-dwelling inhabitants of 48 geo-demographic areas in the Netherlands. The PHARMO registers are linked on a patient level and contain unprecedented accurate and complete information required for the study.

The out patient database contains drug dispensing data in the U-Expo database are encoded according to standards based upon the Z-Index drug database (www.z-index.nl). Therefore, it is possible to identify and classify drug use in time, both on the basis of national and international classification schemes as well as on the basis of individual active ingredients and administration forms. Of each dispensed drug, the Anatomical Therapeutic Chemical (ATC) code, the dispensing date, the prescriber, the prescribed dosage regimen, the dispensed quantity, the cost and the estimated legend duration of use are available.

The hospital pharmacy database comprises hospital pharmacy data collected in a growing number of non-academic hospitals in the Netherlands. Currently, data are collected on patient level for more than one million patients from a representative sample of non-academic hospital pharmacies scattered over the Netherlands. The hospital pharmacy database includes data on in-patient medication orders such as type of drug, dose, and time of administration and duration of use.

The Dutch Medical Register (LMR) is the data source comprising all hospital admissions in the Netherlands (www.prismant.nl). These records include detailed information concerning the primary and secondary discharge diagnoses, diagnostic, surgical and treatment procedures, type and frequency of consultations with medical specialists and dates of hospital admission and discharge. All diagnoses are coded according to the International Classification of Diseases, 9th edition (ICD-9-CM). Currently, data until December 2008 are available.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older; Treatment with either Arixtra or LMWH as initial in-hospital thromboprophylactic agent; At least three months history in the PHARMO RLS database before cohort entry date

Exclusion Criteria:

* Hospitalization for haemorrhage, renal failure or liver failure in the 3 months before cohort entry date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years and older with a primary discharge diagnosis of hip fracture surgery or hospitalization for hip replacement surgery or knee replacement surgery treated with either fondaparinux sodium or LMWH for thrombopropylaxis between January 2003 and September 2008
Sampling Method: Non-Probability Sample
Enrollment: 13442 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Fondaparinux: All dosages of fondaparinux
- Low Molecular Weight Heparins (LMWHs): All dosages of LMWH, including Enoxaparin, Dalteparin, Nadroparin, and Tinzaparin
Period: Overall Study
Arm/Group | Fondaparinux | Low Molecular Weight Heparins (LMWHs)
Started | 1559 | 11883
Completed | 1559 | 11883
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fondaparinux | Low Molecular Weight Heparins (LMWHs) | Total
Number analyzed (Participants) | 1559 | 11883 | 13442
Age, Customized [Number; unit: Participants] — Number of participants falling into the indicated age ranges
  Participants
    18-64 years | 478 | 2962 | 3440
    65-74 years | 568 | 3433 | 4001
    >=75 years | 513 | 5488 | 6001
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1098 | 8280 | 9378
  Male | 461 | 3603 | 4064
Number of participants with the indicated duration of their in-hospital stay [Number; unit: participants]
  0-7 days | 994 | 4826 | 5820
  8-10 days | 428 | 2965 | 3393
  11-14 days | 75 | 1608 | 1683
  >=15 days | 62 | 2484 | 2546
Number of participants hospitalized because of hip surgery and knee surgery [Number; unit: participants]
  Knee surgery | 414 | 3073 | 3487
  Hip surgery | 1145 | 8810 | 9955
Number of participants with the indicated duration of follow-up [Number; unit: participants] — Follow-up includes time in the hospital.
  participants
    1-14 days | 790 | 4331 | 5121
    15-28 days | 477 | 1196 | 1673
    29-42 days | 127 | 2232 | 2359
    >=43 days | 165 | 4124 | 4289
Number of participants with the indicated major risk factors or other key characteristics [Number; unit: participants] — Non-specific non-steroidal anti-inflammatory drugs, ns-NSAIDs; PAU, prior antithrombotic use.
  participants
    PAU: Heparin | 0 | 1 | 1
    PAU: LMWHs | 3 | 42 | 45
    PAU: Vitamin K Antagonist (VKA) | 30 | 351 | 381
    PAU: Fondaparinux | 2 | 0 | 2
    PAU: Multiple agents | 0 | 11 | 11
    Use of platelet inhibitors | 293 | 2610 | 2903
    Use of ns-NSAIDs | 395 | 2717 | 3112
    Hospitalization for hypercoagulable state | 0 | 0 | 0
    Hospitalization for cancer | 7 | 100 | 107
    Hospitalization for thrombocytopenia | 1 | 0 | 1
    Hypertension | 764 | 5645 | 6409
    Cardiovascular disease | 378 | 2923 | 3301
    Hospitalization for cerebrovascular disease | 1 | 30 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Types of Haemorrhages During Hospitalization or Follow-up for Major Orthopaedic Surgery of Lower Limbs (MOSLL)
Description: Haemorrhages during MOSLL hospitalization or follow-up as identified by ICD-9-CM codes were measured. The PHARMO medical record linkage system (RLS), in the Netherlands, is a population-based patient-centric data tracking system that includes high quality/ complete information of patient demographics, drug dispensing, and hospital morbidity records of approximately 2.3 million inhabitants in the Netherlands.
Time Frame: Follow-up continued until the date of first event, death, end of initial therapy, hospital discharge, end of follow-up in PHARMO RLS, or 60 days after discharge, whichever came first
Population: From the PHARMO RLS, all patients >=18 years of age with in-hospital pharmacy data, a primary discharge diagnosis for hip fracture and/or a hospitalization for MOSLL, and follow-up between January 2003 (introduction of Arixtra) and December 2008.
Measure: Number; unit: participants
Arm/Group | Fondaparinux | Low Molecular Weight Heparins (LMWHs)
Number analyzed (Participants) | 1559 | 11883
participants
  Bleeding or hematoma as complication of a surgery | 7 | 10
  Epistaxis | 0 | 3
  Gastrointestinal bleeds | 0 | 9
  Hemarthrosis | 0 | 2
  Intracranial bleeds | 0 | 1
  Urinary tract bleeding | 1 | 1

2. Secondary Outcome: Number of Participants With the Indicated Haemorrhages During Hospitalization for Major Orthopaedic Surgery of Lower Limbs (MOSLL)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux | Low Molecular Weight Heparins (LMWHs)
Number analyzed (Participants) | 1559 | 11883
participants
  Bleeding or hematoma as complication of a surgery | 1 | 0
  Epistaxis | 0 | 1

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing data; thus, no assessments for Serious or Non-serious Adverse Events were performed.
Arm/Group | Fondaparinux | Low Molecular Weight Heparins (LMWHs)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Differences among hospitals in the registration of events (not all events were captured), the presence of policlinical pharmacy, and different drug usage patterns in each hospital did not enable a valid comparison of the risk of haemorrhage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.